CLINICAL TRIAL: NCT02875600
Title: Magnetic Resonance Flow Measurements of Mesenteric Arteries and Veins and Portal Vein With Food Stimulation in Patients Suspected of Chronic Gastro-intestinal Ischemia
Brief Title: Magnetic Resonance Flow Measurements of Mesenteric Arteries and Veins and Portal Vein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Trialbureau radiology, dr, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR flow
Record Dates: First submitted 2016-07-12; First posted 2016-08-23 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Ischemia; Oxygen Deficiency
Keywords: chronic gastro-intestinal ischemia; oxygen deficiency of the gastro-intestinal tract
MeSH Terms: conditions — Ischemia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutri drink (Experimental): MRI flow measurements of mesenterial vessels and portal vein before and after stimulation with nutritional drink
  Interventions: Other: Nutri Drink

INTERVENTIONS:
Other: Nutri Drink — To determine the difference in baseline MR flow measurements and post prandial MR flow measurements between patients diagnosed with CGI and patients not diagnosed with CGI

SUMMARY:
To determine the difference in baseline MR flow measurements and post-prandial MR flow measurements between patients diagnosed with CGI and patients not diagnosed with CGI.

DETAILED DESCRIPTION:
The diagnosis of chronic gastro-intestinal ischemia (CGI) remains a clinical challenge because this diagnosis is difficult to distinguish by the frequent incidence of chronic abdominal pain and asymptomatic stenosis of the mesenteric arteries1. The standard diagnostic work up includes medical history, anamnesis and physical examination, radiological imaging and a functional test as visible light spectroscopy (VLS)2-4 or tonometry5-7. A multidisciplinary team consisting of a gastroenterologist, a vascular surgeon and an interventional radiologist, all specialized in CGI, discusses all patients which results in an expert based consensus diagnosis. Currently, there is no specific test to diagnose CGI. In literature, Magnetic Resonance (MR) techniques are described by which the flow in the mesenteric vessels is measured pre- and post-prandial in healthy volunteers and CGI patients8-12. The flow in the mesenteric vessels increases post-prandial (hyperemia). However, this increase in post-prandial flow compared to pre-prandial appeared less in CGI patients compared to the healthy volunteers. In some CGI patients, even a decrease of the post-prandial compared to pre-prandial flow was seen. We might be able to distinguish patients with CGI from patients without CGI with MR flow measurements with food stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suspected of CGI referred to our hospital for further analysis
2. Age ≥ 18 years
3. Patients who gave informed consent

Exclusion Criteria:

1. Age < 18 years
2. Unable to give informed consent
3. Pregnancy
4. Contra-indications for MRI: a. Metal implants which cannot be removed. E.g. cardiac pacemakers/ICD, aneurysm clips, metal stents, artificial heart valve, cochlea/retinal implants, hearing aids, dentures with magnetic click system or with other metal accessories, tattoos with metallic dye, metal plates/pins/screws of bones, piercings b. Claustrophobia c. Inability to lie still for 1 hour to 1,5 hours
5. Other criteria the physician considers are not compatible with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Determination of difference in baseline MR flow measurements and post prandial MR flow | 2.5 years
  The difference in baseline MR flow measurements and post prandial MR flow measurements between patients diagnosed with CGI and patients not diagnosed with CGI (mL/min/kg)

SECONDARY OUTCOMES:
Wich vessel or combination of vessels differentiate best | 2.5 years
  Which vessel or which combination of vessels best differentiates between patients diagnosed with CGI and patients not diagnosed with CGI by MR flow measurement by computing sensitivity, specificity, predictive positive value and negative predictive value.
The severity of abdominal pain | 20/30/40 minutes
  The severity of abdominal pain in course of time after stimulation with nutritional drink, using the Numeric Pain Intensity scale at baseline and 20, 30 and 40 minutes after nutritional drink
Determination of difference in MR flow measurements before and after treatment for CGI | 2.5 years
  The difference in MR flow measurements of the mesenteric vessels prior to and after treatment in patients diagnosed with CGI with persistent relief of symptoms after treatment (in (mL/min/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ouhlous, md, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmusmc, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No